CLINICAL TRIAL: NCT04437771
Title: Long-Term Follow-up: Phase I/II Clinical Study to Evaluate the Safety and Efficacy of the Infusion of Autologous CD34+ Cells Transduced With a Lentiviral Vector Carrying the FANCA Gene in Patients With Fanconi Anaemia Subtype A: FANCOLEN-I
Brief Title: Long-Term Follow-up of Subjects With Fanconi Anaemia Subtype A Treated With ex Vivo Gene Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RP-L102-0116-LTFU
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Fanconi Anemia Complementation Group A; Fanconi Anemia
Keywords: gene therapy; anaemia; autologous hematopoeitic stem cell transplant; safety; bone marrow failure; genetic diseases; anemia
MeSH Terms: conditions — Fanconi Syndrome; Fanconi Anemia; Anemia; Bone Marrow Failure Disorders; Genetic Diseases, Inborn | interventions — Safety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with Fanconi Anaemia Subtype A (FA-A): Subjects treated with ex vivo lentiviral gene therapy product in FANCOLEN-I trial and agree to participate in this long-term follow-up (LTFU) study
  Interventions: Other: Safety and efficacy assessments

INTERVENTIONS:
Other: Safety and efficacy assessments — Long term disease and gene therapy specific safety evaluations and efficacy assessments

SUMMARY:
This is a long-term safety and efficacy follow-up study for subjects with Fanconi Anaemia Subtype A who have been treated with ex vivo gene therapy on the FANCOLEN-I trial. After completion of the FANCOLEN-I study, eligible subjects will be followed for a total of 15 years post gene therapy treatment. No investigational drug product will be administered during this study.

DETAILED DESCRIPTION:
This long-term follow-up protocol will evaluate the long term safety and efficacy of the infusion of autologous CD34+ cells transduced with lentiviral vector (LV) carrying the FANCA gene.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in the FANCOLEN-I study
2. Treated with gene therapy in the FANCOLEN-I study
3. Able to adhere to the study visit schedule and protocol requirements
4. Provided written informed consent and, as applicable, assent to participate

Exclusion Criteria:

* There are no exclusion criteria for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with Fanconi anemia subtype A who have been treated with ex vivo gene therapy product in FANCOLEN-I study
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2034-10-30 (Estimated); Study Completion 2035-01-30 (Estimated)

PRIMARY OUTCOMES:
Monitor long term safety of patients through blood laboratory evaluations and general health status | 15 years post-drug product infusion
  Evaluate long term safety following infusion of hematopoietic cells transduced with therapeutic lentiviral vector (LV)
Long term genetic correction assessed in bone marrow and blood | 15 years post-drug product infusion
  Determine long term persistence of therapeutic LV in hematopoietic cells in bone marrow and blood
Replication competent lentivirus (RCL) | 15 years post-drug product infusion
  Evaluate RCL in peripheral blood
Insertion site analysis in blood | 15 years post-drug product infusion
  Determine long term clonality
Phenotypic correction | 15 years post-drug product infusion
  Determine phenotypic correction of bone marrow and peripheral blood cells by resistance to DNA-damaging agents
Assessment for Malignancies | 15 years post-drug product infusion
  Monitor for incidence of hematologic malignancies and solid organ tumors
Hematologic stabilization | 15 years post-drug product infusion
  Monitor for long term stability and normalization of blood counts

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Infantil Universitario Niño Jesús (HIUNJ), Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rio P, Zubicaray J, Navarro S, Galvez E, Sanchez-Dominguez R, Nicoletti E, Sebastian E, Rothe M, Pujol R, Bogliolo M, John-Neek P, Bastone AL, Schambach A, Wang W, Schmidt M, Larcher L, Segovia JC, Yanez RM, Alberquilla O, Diez B, Fernandez-Garcia M, Garcia-Garcia L, Ramirez M, Galy A, Lefrere F, Cavazzana M, Leblanc T, Garcia de Andoin N, Lopez-Almaraz R, Catala A, Barquinero J, Rodriguez-Perales S, Rao G, Surralles J, Soulier J, Diaz-de-Heredia C, Schwartz JD, Sevilla J, Bueren JA; FANCOLEN-1 gene therapy investigators. Haematopoietic gene therapy of non-conditioned patients with Fanconi anaemia-A: results from open-label phase 1/2 (FANCOLEN-1) and long-term clinical trials. Lancet. 2025 Dec 21;404(10471):2584-2592. doi: 10.1016/S0140-6736(24)01880-4. Epub 2024 Dec 3. PMID 39642902